CLINICAL TRIAL: NCT02103933
Title: Pilot Study to Evaluate the Knowledge and Understanding on Surgery for Patients With Hysterectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Myong Cheol Lim, Faculty, Center for Uterine Cancer, National Cancer Center, Korea
Other Study IDs: NCC2014-0010
Record Dates: First submitted 2014-03-15; First posted 2014-04-04 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Gynecologic Cancer; Myoma
MeSH Terms: conditions — Myoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the level of knowledge of surgery for women who underwent hysterectomy

ELIGIBILITY:
Inclusion Criteria:

* Women who underwent hysterectomy at National Cancer Center, Korea
* Age > 20 years

Exclusion Criteria:

* The patients who refuse to participate or give consent to the procedure

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who underwent hysterectomy at National Cancer Center, Korea
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Knowledge of hysterectomy | No more than 5 years after hysterectomy
  The questionnaire of hysterectomy knowledge will be conducted by professional experts content validity review.

SECONDARY OUTCOMES:
Decision conflict with hysterectomy | No more than 5 years after hysterectomy
  Decision Conflict Scale(DCS) will be used for decision of conflict with hysterectomy.

OTHER OUTCOMES:
Decision satisfaction with hysterectomy | No more than 5 years after hysterectomy
  Satisfaction with Decision(SWD) will be used for decision of satisfaction with hysterectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Myong Cheol Lim, MD, PhD, Principal Investigator — National Cancer Center, Korea